CLINICAL TRIAL: NCT00551707
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Superiority of CRx-102 Over Each of Its Components When Given to Subjects With Active Rheumatoid Arthritis (RA)
Brief Title: Multicenter Study to Evaluate CRx-102 vs. Each of Its Components to Treat Active Rheumatoid Arthritis
Acronym: MARS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRx-102-007
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis
Keywords: CombinatoRx; CRx-102; Rheumatoid Arthritis; Prednisolone; Dipyridamole; ACR20
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — dipyridamole, prednisolone drug combination; Prednisolone; Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CRx-102 (2.7/180) (Experimental): CRx-102 dose 1 total daily dose during treatment period (days 14-98) 2.7 mg prednisolone plus 180 mg dipyridamole administered as 1.8 mg prednisolone plus 90 mg dipyridamole at 8 AM and 0.9 mg prednisolone plus 90 mg dipyridamole at 1 PM titration dose (days 0-13) 2.7 mg prednisolone plus 90 mg dipyridamole administered as 1.8 mg prednisolone plus 45 mg dipyridamole at 8 AM and 0.9 mg prednisolone plus 45 mg dipyridamole at 1 PM
  Interventions: Drug: CRx-102 (2.7/180)
- CRx-102 (2.7/360) (Experimental): CRx-102 Dose 2 total daily dose during treatment period (days 14-98) 2.7 mg prednisolone plus 360 mg dipyridamole administered as 1.8 mg prednisolone plus 180 mg dipyridamole at 8 AM and 0.9 mg prednisolone plus 180 mg dipyridamole at 1 PM titration dose 1 (days 0-6) 2.7 mg prednisolone plus 90 mg dipyridamole administered as 1.8 mg prednisolone plus 45 mg dipyridamole at 8 AM and 0.9 mg prednisolone plus 45 mg dipyridamole at 1 PM titration dose 2 (days 7-13) 2.7 mg prednisolone plus 180 mg dipyridamole administered as 1.8 mg prednisolone plus 90 mg dipyridamole at 8 AM and 0.9 mg prednisolone plus 90 mg dipyridamole at 1 PM
  Interventions: Drug: CRx-102 (2.7/180); Drug: CRx-102 (2.7/360)
- Prednisolone (Active Comparator): treatment dose ( days 0-98) total daily dose of 2.7 mg prednisolone administered as 1.8 mg prednisolone at 8 AM and 0.9 mg prednisolone at 1 PM
  Interventions: Drug: prednisolone
- Dipyridamole (Active Comparator): total daily dose during treatment period (days 14-98) 360 mg dipyridamole administered as 180 mg dipyridamole at 8 AM and and 180 mg dipyridamole at 1 PM titration dose 1 (days 0-6) 90 mg dipyridamole administered 45 mg dipyridamole at 8 AM and 45 mg dipyridamole at 1 PM titration dose 2 (days 7-13) 180 mg dipyridamole administered as 90 mg dipyridamole at 8 AM and 90 mg dipyridamole at 1 PM
  Interventions: Drug: dipyridamole
- Placebo (Placebo Comparator): placebo administered twice per day at 8 AM and 1 PM
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CRx-102 (2.7/180) — prednisolone 2.7 mg plus dipyridamole 180 mg
  Other Names: prednisolone 2.7 mg plus dipyridamole 180 mg
  Arms: CRx-102 (2.7/180); CRx-102 (2.7/360)
Drug: prednisolone — prednisolone (2.7 mg)
  Arms: Prednisolone
Drug: dipyridamole — dipyridamole 360 mg
  Other Names: dipyridamole 360 mg
  Arms: Dipyridamole
Drug: placebo — placebo
  Arms: Placebo
Drug: CRx-102 (2.7/360) — Prednisolone 2.7 mg plus Dipyridamole 360 mg
  Other Names: Prednisolone 2.7 mg plus Dipyridamole 360 mg
  Arms: CRx-102 (2.7/360)

SUMMARY:
CRx-102 is a synergistic combination drug candidate containing the cardiovascular drug dipyridamole and a very low dose of the glucocorticoid prednisolone. CRx-102 is believed to work through a novel mechanism of action in which dipyridamole selectively amplifies the anti-inflammatory and immunomodulatory activities of the glucocorticoid without replicating the dose-dependent adverse effects. CRx-102 has been associated with clinical benefit in proof of concept studies in subjects with hand Osteoarthritis (OA) and Rheumatoid Arthritis (RA).

In this trial, CRx-102 will be given to subjects with active RA as an add-on therapy to existing stable doses of Disease Modifying Anti-Rheumatic Drugs (DMARDs) including methotrexate (MTX), sulfasalazine, hydroxychloroquine, leflunomide or azathioprine. MTX in combination with other DMARDs (e.g., sulfasalazine or hydroxychloroquine) will be permitted to reflect the current standard of care practices within rheumatology.

DETAILED DESCRIPTION:
The study was discontinued before the enrollment objective was met. Preliminary review of the efficacy dataset revealed that the efficacy dataset was not robust enough to support an extensive formal efficacy analysis as described in the SAP. Therefore, only the CRP values over time and the percent change in C-reactive protein (CRP) values in the As-Treated population were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily give written informed consent
* Subject must be ≥ 18 years of age
* Subject must have RA (ACR criteria)
* Subject must have at least 4 swollen joints and at least 6 tender joints at screening and baseline (28 joint count)
* Subject must have a CRP > Upper Limit of Normal at screening
* Subject must have been on DMARD or DMARD combination (e.g. MTX + hydroxychloroquine) for at least 3 months and be on a stable dose of DMARD(s) for at least 6 weeks prior to screening.
* For MTX subjects: MTX ≥ 7.5 mg weekly (po/sc/im) and willing to take folic acid or folinic acid supplementation
* Subject willing to take concomitant multivitamin or the equivalent of 400 I.U. vitamin D and the equivalent of 1000 mg of elemental calcium daily

Exclusion Criteria:

* History of clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease
* Wheelchair or bed bound
* History of osteoporotic fracture
* History of malignancy within the past 10 years. However, subjects with a history of treated or excised basal cell carcinoma or fewer than 3 squamous cell carcinomas are eligible to participate
* History of lymphoma or chronic leukemia
* Moles or lesions that are currently undiagnosed, but are suspicious for malignancy
* Surgery within the previous 3 months (except for minor dental and cosmetic)
* History of drug or alcohol abuse (as defined by the Investigator)
* History of bleeding disorder
* History of gastrointestinal bleeding within 5 years of screening
* History of severe migraines or headaches
* History of glaucoma
* Active diabetic retinopathy
* Visually compromising cataract
* History of opportunistic infection within the previous 12 months
* Active Tuberculosis (TB)
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening
* Fever or symptomatic viral or bacterial infection within 2 weeks prior to screening
* Positive for Hepatitis C virus (HCV) antibody
* Positive for HBsAg
* Known positive HIV antibody
* Has a history of hypersensitivity to glucocorticoids and/or dipyridamole
* Treatment with oral, intra-articular, intramuscular, or intravenous glucocorticoids within 6 weeks prior to screening; inhaled glucocorticoid is permitted
* Treatment with any tumor necrosis factor-alpha (TNFα) biologic, anakinra or abatacept within 2 months prior to screening
* Treatment with rituximab
* Treatment with another investigational drug 3 months prior to screening
* Treatment with anticoagulants including: dipyridamole, warfarin, clopidogrel, ticlopidine; Acetylsalicylic acid > 150 mg per day
* Treatment with any concomitant medications that have not been at a stable dose for at least 28 days prior to screening
* Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) laboratory values that exceed 1.5 x ULN
* HbA1C value of > 7.0%
* Current enrollment in any other study with investigational drug or device
* Female subject who is pregnant or lactating or of child bearing potential and not using acceptable methods of contraception (birth control pills, barriers or abstinence)
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator or sponsor make the subject unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lee, PhD, Study Director — Zalicus
Locations (48):
- United States (13):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - La Jolla, California
  - Westlake Village, California
  - Palm Harbor, Florida
  - Elizabethtown, Kentucky
  - Haddon Heights, New Jersey
  - Mayfield Village, Ohio
  - Oklahoma City, Oklahoma
  - Dallas, Texas
- Argentina (4):
  - Buenos Aires, Buenos Aires
  - Rosario, Santa Fe Province
  - San Jan
  - San Miguel de Tucumán
- Canada (4):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Hamilton, Ontario
  - Windsor, Ontario
- Estonia (2):
  - Tallinn
  - Tartu
- Hungary (3):
  - Békéscsaba
  - Esztergom
  - Szolnok
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (2):
  - Aguascalientes, Aguascalientes
  - Vallarta Norte, Guadalajara
- Poland (8):
  - Bialystok
  - Elblag
  - Katowice
  - Krakow
  - Lublin
  - Poznan
  - Torun
  - Warsaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Timișoara
- Russia (2):
  - Moscow
  - Saint Petersburg
- Serbia (2):
  - Belgrade
  - Niška Banja
- South Africa (3):
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Worcester, Western Cape

RESULTS

PARTICIPANT FLOW:
Groups:
- CRx-102 (2.7/180): CRx-102 dose 1 2.7 mg prednisolone plus 180 mg dipyridamole
- CRx-102 (2.7/360): Crx-102 (Dose 2)
  2.7 mg prednisolone plus 360 mg dipyridamole
- Prednisolone: prednisolone
  prednisolone: prednisolone (2.7 mg)
- Dipyridamole: dipyridamole
  dipyridamole: dipyridamole (360 mg)
Period: Overall Study
Arm/Group | CRx-102 (2.7/180) | CRx-102 (2.7/360) | Prednisolone | Dipyridamole | Placebo
Started | 4 | 22 | 13 | 8 | 4
Completed | 4 | 16 | 10 | 4 | 3
Not Completed | 0 | 6 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- CRx-102 (2.7/180): Crx-102 (Dose 1) 2.7 mg prednisolone plus 180 mg dipyridamole
- Dipyridamole: dipyridamole
  dipyridamole: dipyridamole (180 mg or 360 mg)
- Total: Total of all reporting groups
Arm/Group | CRx-102 (2.7/180) | CRx-102 (2.7/360) | Prednisolone | Dipyridamole | Placebo | Total
Number analyzed (Participants) | 4 | 22 | 13 | 8 | 4 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (5.50) | 56.2 (11.96) | 55.8 (11.32) | 56.5 (12.76) | 58.8 (9.54) | 56.0 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 18 | 5 | 7 | 3 | 35
  Male | 2 | 4 | 8 | 1 | 1 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline to Day 98 in C-reactive Protein (CRP) Values - As Treated Population
Description: Preliminary review of the efficacy dataset revealed that the efficacy dataset was not robust enough to support an extensive formal efficacy analysis as described in the SAP. Therefore, only the CRP values over time and the percent change in CRP values in the As-Treated population were calculated.
Time Frame: baseline to day 98
Population: As treated population
Measure: Median (Full Range); unit: percentage of change from baseline
Arm/Group | CRx-102 (2.7/180) | CRx-102 (2.7/360) | Prednisolone | Dipyridamole | Placebo
Number analyzed (Participants) | 4 | 16 | 10 | 4 | 3
percentage of change from baseline | -29.90 (18.45) [-36.1 to 3.8] | -40.84 (66.80) [-95.9 to 148.1] | 15.92 (1453.54) [-80.6 to 4617.6] | -33.67 (30.43) [-54.4 to 15.0] | -27.64 [-35.0 to 203.3]

2. Secondary Outcome: To Assess the Superiority of CRx-102 Compared to Prednisolone and Dipyridamole Using American College of Rheumatology Rating Scale (20% or More Improvement; ACR20) Calculated From Baseline to Day 98 in Subjects With Active Rheumatoid Arthritis
Description: as for outcome 1
Time Frame: baseline to day 98
Reporting Status: Not Posted

3. Primary Outcome: Absolute C-reactive Protein (CRP) Values at Day 98 - As Treated Population
Description: as for outcome 1
Time Frame: Day 98
Population: As treated population
Measure: Median (Full Range); unit: mg/L
Groups:
- Dipyridamole: dipyridamole
  dipyridamole: dipyridamole 360 mg
Arm/Group | CRx-102 (2.7/180) | CRx-102 (2.7/360) | Prednisolone | Dipyridamole | Placebo
Number analyzed (Participants) | 4 | 16 | 10 | 4 | 3
mg/L | 12.85 (5.39) [6.6 to 18.9] | 14.25 (15.52) [1.1 to 48.0] | 21.85 (27.10) [1.2 to 80.2] | 16.60 (16.22) [15.9 to 48.8] | 2.68 (4.88) [0.9 to 10.1]

4. Secondary Outcome: To Assess the Efficacy of CRx-102 Compared to Placebo Using ACR 20 Calculated From Baseline to Day 98
Description: as for outcome 1
Time Frame: baseline to 98 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From subject entry into the study (defined as the time at which the informed consent form was signed) to the end of study visit at day 98
Groups:
- CRx-102 (Dose 1): Crx-102 (Dose 1)
  CRx-102: prednisolone + dipyridamole
- CRx-102 (Dose 2): Crx-102 (Dose 2)
  CRx-102: prednisolone + dipyridamole
Arm/Group | CRx-102 (Dose 1) | CRx-102 (Dose 2) | Prednisolone | Dipyridamole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/22 | 0/13 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 10/22 | 2/13 | 4/8 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CRx-102 (Dose 1) (N=4) | CRx-102 (Dose 2) (N=22) | Prednisolone (N=13) | Dipyridamole (N=8) | Placebo (N=4)
Headache (Nervous system disorders) | 0 | 6 | 1 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less